CLINICAL TRIAL: NCT03019302
Title: A Study to Determine the Incidence of Catheter-Related Venous Thrombosis When Using Arrow Peripherally-Inserted Central Catheters With Chlorag+Ard Technology
Brief Title: Arrow Chloragard Peripherally-Inserted Central Catheters (PICC) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Teleflex (Industry)
Collaborators: Arrow International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-07
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Vascular Access Complication; Vascular Access Related Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arrow PICC with Chloragard Technology (Experimental): Arrow Peripherally- Inserted Central Catheters with Chloragard Technology. The application of Chlorag+ard® Technology uses a proprietary process whereby chlorhexidine is chemically bonded to the intra- luminal catheter surfaces from tip to hub, and extra-luminal catheter body.
  Interventions: Device: Arrow PICC with Chloragard Technology

INTERVENTIONS:
Device: Arrow PICC with Chloragard Technology — chlorhexidine is chemically bonded to the intra- luminal catheter surfaces from tip to hub, and extra-luminal catheter body
  Other Names: Chloragard PICC

SUMMARY:
A prospective study evaluating the timing, incidence and relationship of commonly occurring complications related to the use of peripherally-inserted central catheters. All subjects will receive PICC access using the Arrow PICC with Chloragard Technology.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years requiring a PICC for a period of fourteen days or greater (note: maximum study period is 90 days)
* Ability to comply with study requirements inclusive of the follow-up duplex ultrasound procedures and, as applicable, recording of PICC management, interventions and related treatments in the inpatient and outpatient setting in the daily subject diary
* Patients cognitively and physically able to give written consent to participate in the study or patient has a legally authorized representative (LAR) who may give written consent to participate in the study

Exclusion Criteria:

* Previous history of (within 3 months) or current diagnosis of venous thrombosis within the venous tract of the proposed catheter
* History or diagnosis of peripheral or central vein stenosis (on proposed insertion side)
* History or diagnosis of veno-occlusive disease
* History or diagnosis of superior vena cava syndrome
* Known, pre-existing diagnosis of hypercoagulation disorder unrelated to underlying disease
* Previous enrollment in this study
* Currently pregnant or breast feeding
* Previous axillary lymph node dissection on the same side as intended catheter insertion site unless cleared by physician and patient consent
* Skin condition at or within 15 cm of the proposed catheter insertion site, including signs and symptoms of inflammation, rash, crusts, wounds with drainage, sites of intravenous infusion infiltration or extravasation, hematoma, phlebitis and or thrombophlebitis
* Medical, social, and/or psychological problems precluding subject from study participation
* Stage 2, 3 or 4 chronic kidney disease or serum creatinine > 3 mg/dl or Glomerular Filtration Rate (GFR) less than 60 mL per minute per 1.73 m2 unless cleared by a nephrologist for participation
* Known allergy or sensitivity to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic and asymptomatic catheter-related venous thrombosis (CVRT) | within maximum 90 days dwell
Incidence of catheter occlusion | within maximum 90 days dwell
Incidence of catheter-related bloodstream infections | within maximum 90 days dwell

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Detroit Medical Center, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No